CLINICAL TRIAL: NCT05977283
Title: An Observational Follow-up Study to Describe Treatment Patterns and Outcomes in Hepatitis B Patients With HBsAg Decline in Past 6 Months
Brief Title: HBsAg Declined Patients Follow-up Study
Status: Recruiting | Type: Observational
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2022-260
Record Dates: First submitted 2022-11-29; First posted 2023-08-04 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Hepatitis B; Hepatitis B, Chronic
Keywords: chronic hepatitis b; HBsAg; functional cure
MeSH Terms: conditions — Hepatitis B; Hepatitis B, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Participants will be asked to store a certain amount of blood samples in site during study visit for future HBV markers, host immunity or other related tests. The retained remaining samples from previous tests before this follow-up study may also be used for HBV related exploratory research after patient informed consent.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to prospectively follow chronic hepatitis B patients who had HBsAg decline in the past 12 months prior to screening. The main question it aims to answer are:

- Describe treatment pattern and its impact on HBsAg loss in hepatitis B patients who had HBsAg decline in past 12 months due to any reason (with or without new molecular entities therapy).

Participants will be followed up for 36 months after enrollment and may be extended upon expiration according to study objectives.

DETAILED DESCRIPTION:
This study is a retrospective and prospective follow-up study for participants who had HBsAg decline in past 6 months due to any reason (with or without new molecular entities therapy). The follow-up period will be 3 years (36 months after enrollment) and may be extended upon expiration according to study objectives. Patients are treated or untreated based on current clinical practice guidelines, and every medical decision and course of treatment will reflect exclusively the decision of the treating physician in a routine clinical situation. The conduct of this non-interventional follow-up study and its documentation procedures will not affect the routine treatment of the subjects. It is only requested that any medical decisions, procedures and data during this study be documented in the electronic case report/record form (eCRF) according to the study protocol as available from routine medical care. Diagnostic testing and monitoring procedures are exclusively based on the decision of the treating physician.

In general, patients with hepatitis B should be monitored at least twice a year (every 6 months), every 12 weeks during NUC therapy and every 2 to 4 weeks during interferon-α therapy in accordance with clinical needs (Table 3-1 and Table 3-2). For patients had HBsAg decline in past 6 months due to new molecular entities therapy, The baseline of this follow-up study is the time when NME discontinued (within 28 days of the last does of NME or within 2 half-life period of the NME). For patients had HBsAg decline in past 6 months without new molecular entities therapy, the baseline should be the time of enrolling in the study. The time of enrolling in this study may be posterior or equal to baseline, which is not necessarily the baseline of this study. The visit window period is ±28 days for patients with NUC therapy and ±7 days for patients with interferon-α therapy. Follow-up study visit data can be collected retrospectively if it has been performed before entry of this study.

Medical decisions, procedures and data before this follow-up study will also be documented if available. Participants will be asked to store a certain amount of blood samples in site during study visit for future HBV markers, host immunity or other related tests. The retained remaining samples from previous tests before this follow-up study may also be used for HBV related exploratory research after patient informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have HBsAg decline ≥0.5 log10 IU/mL in past 12 months prior to screening due to any reason (with or without new molecular entities therapy). Among the enrolled subjects, 70% must have HBsAg decline ≥1 log10 IU/mL or actual values ≤3 log10 IU/mL.
* Able and willing to provide written informed consent and to comply with the study protocol according to International Council for Harmonization (ICH) and local regulations.

Exclusion Criteria:

* Any condition which, in the opinion of the investigator, contraindicates their participant in this study.
* Participants who are currently participating in interventional clinical study exploring HBV treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants must have HBsAg decline ≥0.5 log10 IU/mL in past 12 months prior to screening due to any reason (with or without new molecular entities therapy). Among the enrolled subjects, 70% must have HBsAg decline ≥1 log10 IU/mL or actual values ≤3 log10 IU/mL.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-05-11 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with HBsAg loss (<0.05 IU/ml) at 12 months | at week 48
  Describe treatment pattern and its impact on HBsAg loss of the included patients (with or without new molecular entities therapy) by the proportion of participants with HBsAg loss at week 48.

SECONDARY OUTCOMES:
Proportion of participants with HBsAg loss or HBsAg seroconversion. | at week 48, 96 and 144
  HBsAg loss / seroconversion at each study visit
Change from baseline in quantitative HBsAg levels over time | at week 48, 96 and 144
  including but not limited to actual values and changes from Baseline (Pre-treatment, 6 month prior to screening, and the beginning of follow-up study) at week 48, 96 and 144 in HBsAg, HBV DNA, HBeAg, HBcrAg, HBV RNA level
Change from baseline in quantitative anti-HBs levels over time | at week 48, 96 and 144
  Describe the development of anti-HBs over time for hepatitis B patients with HBsAg decline in past 6 months due to any reason (with or without new molecular entities therapy)
Incidence of liver cirrhosis, hepatocellular carcinoma, other HBV complications and mortality, at each study visit | at week 48, 96 and 144
  The incidence of de novo liver cirrhosis, hepatocellular carcinoma, other HBV complications and mortality
The change of Health-related quality-of-life (HRQoL) over time | at week 48, 96 and 144
  evaluated the risk factors on the progression of CHB, by the available data

CONTACTS AND LOCATIONS:
Overall Officials: jinlin hou, Master, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] BLUMBERG BS, ALTER HJ, VISNICH S. A "NEW" ANTIGEN IN LEUKEMIA SERA. JAMA. 1965 Feb 15;191:541-6. doi: 10.1001/jama.1965.03080070025007. No abstract available. PMID 14239025
- [Background] European Association for the Study of the Liver. EASL 2017 Clinical Practice Guidelines on the management of hepatitis B virus infection. J Hepatol. 2017 Aug;67(2):370-398. doi: 10.1016/j.jhep.2017.03.021. Epub 2017 Apr 18. PMID 28427875
- [Background] Brunetto MR. A new role for an old marker, HBsAg. J Hepatol. 2010 Apr;52(4):475-7. doi: 10.1016/j.jhep.2009.12.020. Epub 2010 Jan 30. No abstract available. PMID 20185190
- [Background] Chan HL, Thompson A, Martinot-Peignoux M, Piratvisuth T, Cornberg M, Brunetto MR, Tillmann HL, Kao JH, Jia JD, Wedemeyer H, Locarnini S, Janssen HL, Marcellin P. Hepatitis B surface antigen quantification: why and how to use it in 2011 - a core group report. J Hepatol. 2011 Nov;55(5):1121-31. doi: 10.1016/j.jhep.2011.06.006. Epub 2011 Jun 28. PMID 21718667
- [Background] - Lau G K K, Marcellin P, Brunetto M, et al. 917 on-treatment monitoring of HBsAg levels to predict response to peginterferon alfa-2a in patients with HBeAg-positive chronic hepatitis B[J]. Journal of Hepatology, 2009, 50, Supplement 1(0): S333